CLINICAL TRIAL: NCT07284381
Title: A Multicenter, Double-masked, Randomized Study to Compare the Efficacy and Safety of the ABBV-444 Tear Formulation With REFRESH OPTIVE® Unit Dose in Patients With Dry Eye Disease
Brief Title: A Clinical Study to Evaluate the Effect and Side Effect of a New Artificial Tear Formulation (ABBV-444) Compared to Refresh Optive Unit Dose in Adult Participants With Dry Eye Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M23-730
Record Dates: First submitted 2025-12-08; First posted 2025-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye Disease; ABBV-444
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABBV-444 (Experimental): Participant will receive ABBV-444 as needed but at least twice a day for 90 days.
  Interventions: Drug: ABBV-444
- REFRESH OPTIVE UD (Active Comparator): Participant will receive REFRESH PLUS as needed but at least twice a day for 90 days. (Refresh Plus is the run-in medication for 7-10 days before study treatment assignment)
  Interventions: Drug: REFRESH OPTIVE UD

INTERVENTIONS:
Drug: ABBV-444 — Topical eye drop
  Arms: ABBV-444
Drug: REFRESH OPTIVE UD — Topical eye drop
  Arms: REFRESH OPTIVE UD

SUMMARY:
Dry Eye Disease (DED) refers to a long-term condition that happens when there is not enough lubrication in your eyes. This can happen when your eye cannot make enough tears or if you make poor-quality tears. The purpose of this study is to compare the efficacy and safety of a new artificial tear formulation (ABBV-444) with Refresh Optive UD for 90 days in participants with Dry Eye Disease (DED.

ABBV-444 is being developed for the treatment of Dry Eye Disease (DED). Participants will be placed into 1 of 2 treatment arms. Each group receives different treatment. Adult participants diagnosed with dry eye disease will be enrolled. Around 250 participants will be enrolled in the study at approximately 20 sites across the US

In this study, participants first complete a 7-day run-in period using REFRESH PLUS® eye drops. Those eligible are then randomized to receive ABBV-444 eye drops or REFRESH OPTIVE® Unit Dose eye drops. Participants in both arms will receive treatment for a 90-day treatment period.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend multiple required study visits during the study at the study site. The effect of the treatment will be checked by medical assessments and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Ocular Surface Disease Index (OSDI) score of ≥ 28 and ≤ 65 (based upon a 0 to 100 scale) at Screening. (Day -7) and an OSDI score of ≥ 18 and ≤ 65 (based upon a 0 to 100 scale) at Baseline (Day 1).
* Three consecutive tear breakup time (TBUT) tests of ≤ 10 seconds in at least 1 eye at both the Screening (Day -7) and Baseline (Day 1) Visits.
* Grade 1 to 4 (modified National Eye Institute [NEI] Grid, score range = 0 to 5) staining in at least 1 area of the cornea (5 areas examined) or conjunctiva (6 areas examined) that is related to dry eye in at least 1 eye at both Screening (Day -7) and Baseline (Day 1).
* Have used an artificial tear product for dry eye disease (DED) within 6 months of Screening (Day -7) Visit.

Exclusion Criteria:

* Participant has uncontrolled severe systemic disease that, in the assessment of the investigator, would put safety of the subject at risk through participation, or which would prevent or confound protocol-specified assessments (e.g., hypertension and diabetes, Sjögren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, immunodeficiency disease, etc.).
* Participant has worn contact lenses in the last 90 days prior to the Screening (Day -7) Visit and/or participant anticipates contact lens wear during the study.
* Any scheduled or planned systemic surgery or procedure during the study, which in the investigator's opinion, may impact the participant's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Ocular Surface Disease Index (OSDI) Score | Baseline to Day 90
  The OSDI is a 12-question survey for patients to document their dry eye disease symptoms. The OSDI consists of a 5- point scale (0=none of the time to 4=all of the time), with higher scores representing worse symptoms. The scores are totaled over the 12 questions and converted to a score of 0-100 (0=no symptom to 100=worst symptom). A negative number change from baseline represents an improvement.
Number of Participants with Adverse Events (AEs) | Baseline to Day 90
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from Baseline in Total Ocular Surface Staining Score (OS Staining) (modified NEI Grid, with fluorescein for cornea; and lissamine green for conjunctiva) | Baseline to Day 90
  Corneal staining will be evaluated in each eye at all visits and will be graded 2 minutes after instillation of the fluorescein, during which time TBUT is measured. Grade staining independently approximately 3 minutes in the 5 zones of the cornea (1 through 5) as shown below based upon a 6-point scale (0,
  1, 2, 3, 4, 5) for a maximum grade of 5 in each of the 5 zones (or a total maximal score of 25 for each eye).
Change from Baseline in Tear Breakup Time (TBUT) with Fluorescein | Baseline to Day 90
  The TBUT will be determined during the approximately 3 minutes wait for corneal staining using fluorescein strips moistened with saline drops applied to the treatment area. Participants will be asked to blink normally 2 to 3 times to evenly spread the fluorescein. Then, they will be asked to not blink for as long as they can. As soon as they start holding the blink, the timing with the stopwatch will begin. The stopwatch is stopped on the first occurrence of true tear break-up, not just local thinning or tear film irregularity

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- United States (11):
  - Arizona Eye Center - West Ray Road /ID# 267993, Chandler, Arizona
  - Canyon City Eyecare /ID# 267948, Azusa, California
  - Global Research Management /ID# 267980, Glendale, California
  - Lakeside Vision Center /ID# 268544, Irvine, California
  - Eye Research Foundation /ID# 267931, Newport Beach, California
  - Lee Shettle Eye and Hearing /ID# 268118, Largo, Florida
  - Clayton Eye Center /ID# 268097, Morrow, Georgia
  - Core Inc /ID# 267946, Shelby, North Carolina
  - Scott and Christie and Associates /ID# 268119, Cranberry Township, Pennsylvania
  - Total Eye Care - Memphis /ID# 268327, Memphis, Tennessee
  - Piedmont Eye Center /ID# 267929, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-730